CLINICAL TRIAL: NCT06199518
Title: Comparison of Laparoscopic Ureterolithotomy, Retrograde Flexible Ureteroscopy, and Mini- Percutaneous Antegrade Ureteroscopic Lithotripsy for the Management of Large Proximal Ureteral Stones (1.5-2 cm): A Prospective Randomized Trial.
Brief Title: Minimally Invasive Techniques for Treating Large Proximal Ureteral Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Zoeir, faculty of medicine, Tanta, ElGeish street, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34619/4/21
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Endourology

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP(A):transperitoneal laparoscopic ureterolithotomy (T-LUL) (Active Comparator): extraction of proximal ureteral stones by laparoscopic surgery via transperitoneal approach
  Interventions: Procedure: transperitoneal laparoscopic ureterolithotomy (T-LUL)/ retrograde flexible ureteroscopy (R-URS) /Antegrade mini-percutaneous flexible ureteroscopy (A-URS)
- GROUP (B):retrograde flexible ureteroscopy (R-URS) (Active Comparator): laser lithotripsy of proximal ureteral stones via flexible ureteroscopy retrograde
  Interventions: Procedure: transperitoneal laparoscopic ureterolithotomy (T-LUL)/ retrograde flexible ureteroscopy (R-URS) /Antegrade mini-percutaneous flexible ureteroscopy (A-URS)
- GROUP (C):Antegrade mini-percutaneous flexible ureteroscopy (A-URS) (Active Comparator): laser lithotripsy of proximal ureteral stones via percutanous antegrade flexible ureteroscopy
  Interventions: Procedure: transperitoneal laparoscopic ureterolithotomy (T-LUL)/ retrograde flexible ureteroscopy (R-URS) /Antegrade mini-percutaneous flexible ureteroscopy (A-URS)

INTERVENTIONS:
Procedure: transperitoneal laparoscopic ureterolithotomy (T-LUL)/ retrograde flexible ureteroscopy (R-URS) /Antegrade mini-percutaneous flexible ureteroscopy (A-URS) — extraction or fragmentation of large proximal ureteral stones via different minimally invasive procedures

SUMMARY:
a prospective comparative study designed to compare the outcomes of transperitoneal Laparoscopic ureterolithotomy (T-LUL), mini-percutaneous antegrade ureteroscopy (A-URS) and retrograde ureteroscopy (R-URS) in treating patients with LPUS (15-20 mm). the following parameters were assessed and compared (demographic data and stones characteristics, Stone free rate and complications)

DETAILED DESCRIPTION:
we aimed in the current study to comprehensively evaluate and to compare the outcome of transperitoneal laparoscopic ureterolithtomy, retrograde ureteroscopy and mini-percutaneous antegrade ureteroscopy for management of large proximal ureteric stone (15 -20 mm) with regards to; operative time, stone free rate, success rate, hospital stay and complications.

A total of 105 participants were enrolled in the trial between April 2021 and June 2023 to accomplish this. Inclusion criteria for this study included patients who had a single proximal Ureteral stone (between the pelvi ureteric junction and the upper border of the sacroiliac joint) measuring 15-20 mm in diameter.

Patients were randomly allocated to receive either TPLU, RURS, or Minin-perc Antegrade URS, with a 1:1:1 allocation ratio. After providing informed permission, the patients were randomly assigned to one of three groups: Group I (35 patients treated with TPLU), Group II (35 patients treated with RURS), and Group III (35 patients not treated with either TPLU or RURS) (Included 35 patients who were treated by Mini-perc Antegrade URS)

ELIGIBILITY:
Inclusion Criteria:

* Adults patients
* large proximal ureteral stones(1.5-2 cm)

Exclusion Criteria:

* larger stones
* multiple stones
* bleeding tendency
* active UTI
* distal stricture

Ages: 26 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
stone free rate (SFR) | immediate (initial SFR ) and 1 -month later (final SFR)
  SFR is defined as no residual stones or fragments ≤ 4 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Urolgy Departement, Faculty of Medicine, Tanta University, Tanta, Outside U.S./Canada, Egypt